CLINICAL TRIAL: NCT04034212
Title: Singing for Health: Improving Experiences of Lung Disease (SHIELD Trial)
Acronym: SHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS Project ID: 259170; 19IC5000 (Other: Imperial College London)
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Singing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking of participants not possible due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Singing for Lung Health group (Experimental): Once weekly attendance at a Singing for Lung Health group for 12 weeks.
  Interventions: Other: Singing for Lung Health group attendance
- Usual Care group (No Intervention): Usual care group, participants given advice on physical activity while continuing with usual care.

INTERVENTIONS:
Other: Singing for Lung Health group attendance — Singing for Lung Health is a group singing intervention designed for people with chronic lung diseases. Participants would attend weekly sessions lasting 1 hour.
  Arms: Singing for Lung Health group

SUMMARY:
A randomised clinical trial to assess the impact of group singing on health for people with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Singing for lung health (SLH) is a novel approach intended to improve the health status of people with respiratory disease. In group sessions, a trained singing leader teaches vocal techniques, which improve breathing control and posture, in the context of an enjoyable non-disease related activity. Initial pilot studies and qualitative work have established the concept that SLH can produce physical, psychological and social benefits. A properly conducted efficacy study is needed before larger scale trials, addressing impacts over a longer term and effect on health resource utilisation, can be undertaken.

DESIGN: An assessor blind, parallel group, randomised controlled trial, to assess the effects of SLH compared to usual care on health status. The investigator will also evaluate the impact on physical activity, physical performance, and breathlessness perception to investigate the mechanisms involved.

Research question and outcome measures:

The primary outcome will be change in health status, assessed using the Short Form 36 tool (SF-36), comparing SLH and control arms.

Additional endpoints will be: the COPD assessment test score (CAT), the MRC dyspnoea score, Dyspnoea-12, Activities-specific Balance Confidence scale (ABC scale).

For psychological health, anxiety will be assessed using the GAD-7 and depression using the PHQ-9.

Physical activity will be assessed using the cPPAC PROactive physical activity in COPD tool (a combination of questionnaire and actigraphy). Physical capacity using the six-minute walk test, and physical performance using the short physical performance battery.

Assessments: At an initial baseline assessment a structured clinical history will take place and the diagnosis confirmed by spirometry. The outcomes outlined above will be recorded at baseline and then after 12 weeks.

POPULATION: Adult patients with COPD will be recruited from primary and secondary care as well as through advertising. Diagnosis will be based on clinical history, confirmed by spirometry and a history of smoking. Participants in the active arm will attend once weekly SLH groups for 12 weeks. The comparison arm will receive usual care. Randomization will be stratified by prior participation in pulmonary rehabilitation and by MRC dyspnoea score, to ensure groups are matched.

SAMPLE SIZE Sample size: Based on pilot data, where the standard deviation (SD) for change in SF-36 was 15 points, to identify a clinically relevant 10 point difference in SF-36 responses at a 0.05 level of significance with a 90% power would require 48 patients in each treatment arm. Allowing for 20% dropout the investigator will therefore recruit 120 patients.

Primary analysis will be on an intention to treat basis. Change in parameters will be assessed comparing SLH/control using Generalised Linear Models to estimate treatment effects. In order to better understand changes in the SF-36 "anchor measure", the investigator will relate this to changes in measures of breathlessness, physical activity, capacity and performance.

An additional responder analysis will compare the proportion in each treatment arm achieving a clinically important (10%) improvement in SF-36.

Addendum: Due to the COVID-19 pandemic an it became inappropriate to continue delivering group singing sessions in person, so the first group of participants is to complete their 12 weeks of intervention using online delivered sessions. This relates the first group of 18 participants had been recruited, randomised, baseline assessments completed and begun the intervention. Their follow-assessments will be posted to participants for them to complete at home. All assessment measures will be the same as originally stated, however the 6MWT and SPPB require clinical supervision, so will not be completed. The results from this group will be reported separately to the rest of the study who will complete the original protocol when the situation with COVID-19 has improved, and it is safe for participants to do so. An appropriate amendment to ethical approval has been made. Data from the control group may also be reported separately, being of interest in itself, as a natural experiment regarding the impact of social distancing and shielding measures on people with COPD. Again, the variables assessed will not change.

Addendum 2: Due to the ongoing COVID-19 pandemic, the study will continue to be conducted remotely, as described above, with online delivery of the singing intervention and remotely collected outcome measures. Most recent clinical spirometry will be used for COPD diagnosis confirmation. Due to no longer being able to conduct the object assessments of physical performance mean daily step count will also be reported as a secondary outcome measure. For clarification, the exclusion criteria of previous participation in Singing For Lung health, refers to no participation in the last year. Appropriate amendments to the ethical approval have been made.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stable COPD

Exclusion Criteria:

* Pulmonary rehabilitation less than 4 months ago
* Unable to take part in singing sessions due to comorbidity (e.g. life limiting illness, cognitive impairment)
* Previous participation in SLH classes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Short Form 36 tool (SF-36) | At baseline, then repeated after 12 weeks.
  A well-established, supervised, self-completion health status questionnaire. This consists of eight sections for which a score of 0 to 100 is created, with 0 being maximum disability and 100 equivalent to no disability.

SECONDARY OUTCOMES:
Changes in COPD assessment test (CAT) | At baseline, then repeated after 12 weeks.
  a disease specific health status measure. This includes 8 items, scored 0-5 with a possible score from 0 (best) to 40 (worst).
Changes in Generalised Anxiety Disorder Assessment (GAD-7) | At baseline, then repeated after 12 weeks.
  Self-administered questionnaire to assess for symptoms, and severity, of anxiety. Includes seven questions scored from 0 to 3, giving a total score out of 21. Lower scores indicate less symptoms of anxiety.
Changes in Patient Health Questionnaire 9 (PHQ-9) | At baseline, then repeated after 12 weeks.
  Self-administered questionnaire to assess for symptoms, and severity, of depression. Includes nine questions scored from 0 to 3, giving a total score out of 27. Lower scores indicate less symptoms of depression.
Changes in Dyspnoea-12 questionnaire | At baseline, then repeated after 12 weeks.
  Assessment of dyspnoea. Includes 12 descriptors scored from 0 to 3, giving a total score of 36. Lower scores indicate less severe dyspnoea.
Changes in Six-minute walk test | At baseline, then repeated after 12 weeks.
  Distance walked in 6 minutes. Tests exercise capacity. To be performed in accordance with ATS/ERS guidelines including a practice walk.
Changes in PROactive physical activity in COPD tool (cPPAC) | At baseline, then repeated after 12 weeks.
  This involves a one week recall questionnaire and McRoberts MoveMonitor device physical activity monitor.
Changes in Activities-specific Balance Confidence scale | At baseline, then repeated after 12 weeks.
  Balance confidence during activities of daily living, assessed using self-reported questionnaire. 16 item scale which gives a total balance confidence score of 0 to 100. Lower scores indicate less confidence.
Changes in Short Physical Performance Battery (SPPB) | At baseline, then repeated after 12 weeks.
  Physical performance evaluated using the SPPB (instrumented with the McRoberts fixed-body sensor MoveTest device). Consists of 4 performance tasks (balance, walk speed and sit-to-stand) scored from 0 to 4, giving a total score out of 12 for SPPB.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hopkinson, Study Chair — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philip KEJ, Buttery SC, Bowen S, Lewis A, Jeffery E, Alghamdi SM, Williams P, Alasmari AM, Alsulayyim AS, Orton CM, Conway F, Chan L, Vijayakumar B, Tana A, Tonkin J, Perkins A, Garner JL, Srikanthan K, Sadaka A, Pavitt MJ, Banya W, Lound A, Elkin S, Polkey MI, Man WD, Lewis K, Cave P, Fancourt D, Hopkinson NS. Singing for lung health in COPD: a multicentre randomised controlled trial of online delivery. BMJ Open Respir Res. 2024 May 2;11(1):e002365. doi: 10.1136/bmjresp-2024-002365. PMID 38697677